CLINICAL TRIAL: NCT02158689
Title: Comparison of Treatment Modalities in Poor Responders Undergoing IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ercan Bastu (Other)
Responsible Party: Sponsor-Investigator, Ercan Bastu, Associate Professor of Obstetrics and Gynecology, Istanbul University
Organization: Istanbul University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10017
Record Dates: First submitted 2014-05-27; First posted 2014-06-09 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Poor Responders
Keywords: Poor responders; letrozole; human menopausal gonadotropin
MeSH Terms: interventions — Letrozole; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- human menopausal gonadotropin (hMG) (Active Comparator): hMG at a dose of 300 IU/day will be initiated on the second or third day of spontaneous menstruation and continued until the day of ovulation triggering. Ovulation triggering will be performed with the administration of 10000 IU of human chorionic gonadotropin (hCG) as soon as two-three follicles of 17 mm diameter will be observed by transvaginal ultrasound.
  Interventions: Drug: human menopausal gonadotropin (hMG)
- Letrozole (Active Comparator): Letrozole (Femara; Novartis, East Hanover, NJ) at a dose of 5 mg/day will be initiated on the second or third day of spontaneous menstruation and continued for 5 days. Again on the second or third day of spontaneous menstruation, 150 IU of hMG will be started until the day of ovulation triggering. Ovulation triggering will be performed with the administration of 10000 IU of hCG as soon as two-three follicles of 17 mm diameter will be observed by transvaginal ultrasound.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole
  Other Names: Femara
  Arms: Letrozole
Drug: human menopausal gonadotropin (hMG)
  Arms: human menopausal gonadotropin (hMG)

SUMMARY:
The accurate identification and efficient management of poor responders remains one of the most enigmatic challenges in assisted reproductive technology (ART). The investigators study will compare the letrozole/antagonist protocol to the hMG/antagonist protocol in women who poor responders.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be considered eligible if they are poor ovarian responders according to the Bologna criteria (Ferraretti et al., 2011).
* Two out of three of the following criteria are essential in order to classify a patient as poor ovarian responder:

  * advanced maternal age (≥40 years) or any other risk factor for poor ovarian response;
  * a poor ovarian response (≤3 oocytes with a conventional stimulation protocol); or
  * an abnormal ovarian reserve test (antral follicle count, <7 follicles or anti-Mullerian hormone, <1.1 ng/ml).

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | up to 2 weeks
  The primary outcome measure will be the ongoing pregnancy rate (>12 weeks' gestation) per started cycle.

SECONDARY OUTCOMES:
Cancellation Rate | up to one month
  One of the secondary outcome measures will be cancellation rate.
Number of oocytes retrieved | up to one month
  One of the secondary outcome measures will be number of oocytes retrieved.
Number of transferable embryos | up to one month
  One of the secondary outcome measures will be number of transferable embryos.
Implantation rate | up to 2 weeks
  One of the secondary outcome measures will be implantation rates.
Clinical pregnancy rate | up to 2 weeks
  One of the secondary outcome measures will be clinical pregnancy rates.

CONTACTS AND LOCATIONS:
Overall Officials: Harika Yumru, M.D., Principal Investigator — Istanbul University School of Medicine; Hasan F Buyru, M.D. Prof., Study Chair — Istanbul University School of Medicine; Ercan Bastu, M.D., Study Director — Istanbul University School of Medicine
Locations (1):
- Department of Obstetrics and Gynecology, Istanbul University School of Medicine, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041